CLINICAL TRIAL: NCT06254885
Title: Clinical and Radiographic Evaluation of Equicrestal and Subcrestal Positioning of a Tissue Level Implant With Convergent Transmucosal Profile - Randomized Clinical Trial
Brief Title: Insertion Protocol of Convergent Transmucosal Design Implants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Nicola Alberto Valente, DDS, MS, PhD, Assistant Professor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PramaNAV
Record Dates: First submitted 2024-01-17; First posted 2024-02-12 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Implant Site Reaction
Keywords: Peri-implant mucosa; Peri-implant bone; Transmucosal profile

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sub-crestal (Experimental): Implants will be placed 1mm under the bone crest level
  Interventions: Procedure: Sub-crestal Implant placement
- Equi-crestal (Active Comparator): Implants will be placed at the bone crest level
  Interventions: Procedure: Equi-crestal Implant placement

INTERVENTIONS:
Procedure: Equi-crestal Implant placement — A site will be prepared through consecutive drillings on an edentulous space of the osseous ridge after flap elevation. Then a titanium fixture will be screwed that will serve, after osseointegration, to carry a dental prosthesis. The implant will be screwed until the shoulder (upper marginal part of the implant) is exactly at the same level as the bone of the maxillary/mandibular edentulous crest.
  Arms: Equi-crestal
Procedure: Sub-crestal Implant placement — A site will be prepared through consecutive drillings on an edentulous space of the osseous ridge after flap elevation. Then a titanium fixture will be screwed that will serve, after osseointegration, to carry a dental prosthesis. The implant will be screwed until the shoulder (upper marginal part of the implant) is 1mm below the level of the bone crest.
  Arms: Sub-crestal

SUMMARY:
The aim of this randomized clinical study is the evaluation of the peri-implant mucosal tissues and the marginal bone level, after positioning the transition shoulder from the intraosseous to the transmucosal portion, with an equicrestal position (at the level of the bone crest) or subcrestal (under the bone crest level).

DETAILED DESCRIPTION:
The primary outcomes will be the measurement of the marginal bone level (MBL) at various time intervals and the evaluation of the soft tissues according to a score defined as Pink Esthetic Score (PES). Secondary outcomes will be plaque index (PI); the bleeding index (BI), biological complications (peri-implant mucositis, peri-implantitis, abscesses), implant failure, prosthetic complications (chipping, fractures) and prosthetic failure.

The subjects recruited for the study will be those belonging to the oral surgery department of the San Giovanni di Dio Hospital in Cagliari.

Each patient will receive only one implant or, in any case, only one implant per patient will be included in the analysis. A random sequence will be generated via Randomization.com, useful for assigning patients into the equicrestal and subcrestal implant placement groups.

All patients will undergo the same preoperative, intraoperative and postoperative procedures.

Preoperative procedures An intraoral radiograph of the edentulous site will be performed. Upper and lower alginate impressions will be made on each patient for planning and fabrication of surgical guides, all patients will receive rigorous oral hygiene and instructions will be provided to improve and maintain home oral hygiene.

Intraoperative procedures After local anesthesia of the site to be operated on, a full thickness mucoperiosteal flap will be elevated, after lifting the flap the implant site will be prepared according to the manufacturer's protocol. Before implant placement, the sealed envelope will be opened for random assignment of the patient to one of the two groups. The implant will therefore be positioned, depending on the assignment group, in an equicrestal or subcrestal position, in the latter case a further step with the last preparation drill will be performed to deepen the site.

The flap will be sutured after placement of the healing screw and specific hygiene instructions for the healing site will be given to the patient. The appropriate analgesic and antibiotic therapy will be prescribed.

An intraoral x-ray will be performed in a standardized and repeatable manner to assess bone levels.

The patient will be followed following the following follow-up scheme, reserving the right to recall the patients involved even at longer time intervals to evaluate the aforementioned outcomes also in the medium (24 months) and long (5-10 years) term.

1. week: healing check
2. weeks: healing check and suture removal

1 month: healing check 3 months: prosthesis and intraoral x-ray, measurement of soft tissue parameters via PES after positioning of the prosthetic crown 6 months: intraoral x-ray and PES 12 months: intraoral x-ray and PES The marginal bone level will be measured using ImageJ software (NIH freeware) on the distal and mesial aspects of each implant at each time point where it is foreseen.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Absence of periodontal disease
* Full mouth plaque score and full mouth bleeding score less than or equal to 25%
* Sufficient bone height and width to place an implant in a prosthetically guided position without performing bone grafting procedures
* Stable occlusion

Exclusion Criteria:

* Smokers (more than 10 cigarettes a day)
* Medical conditions that contraindicate implant surgery
* Pregnant and breastfeeding patients
* Patients with a history of therapy with bisphosphonates or biologics
* Patients undergoing chemotherapy or radiation therapy of the head and neck
* Decompensated diabetes
* Severe bruxism
* Poor oral hygiene or uncooperative patients (incomplete data collection or failure to attend scheduled check-up appointments)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Peri-implant mucosa health and condition in terms of Pink Esthetic Score (PES). | 6-12 months
  The PES (Pink Esthetic Score) is a score that evaluates the appearance of the peri-implant soft tissues which examines various parameters giving a value from 0 (worst) to 2 (best) each. (1. the presence/absence of the interproximal papilla both mesial and distal (0=absent, 2=complete); 2. the festooning of the gingival margin in correspondence with the implant (0=unnatural, 2=natural); 3. the position of the gingival margin (0=major discrepancy from reference tooth, 2=no discrepancy); 4. the color of the soft tissues (0=obvious difference from reference tooth, 2=no difference); 5. the appearance (texture) of the soft tissues (0=obvious difference from reference tooth, 2=no difference); 6. defects of the alveolar process (0=obvious deficiency, 2=no deficiency)).
Peri-implant mucosa health and condition in terms of Plaque Index (PI). | 6-12 months
  The Plaque Index (PI) will be calculated. A value of 0 will be assigned if supragingival plaque is not visible, a value of 1 if visible.
Peri-implant mucosa health and condition in terms of Bleeding Index (BI) | 6-12 months
  The Bleeding Index will be calculated on the sites where the periodontal probing will be carried out, a procedure for measuring the depth of the gingival sulcus on 6 sites per tooth (mesial, central, distal, both vestibular and lingual) with a periodontal probe. A value of 0 will be given if there is no bleeding and 1 if the site bleeds within 30 seconds
Peri-implant bone health and condition in terms of change in marginal bone level (MBL) | 6-12 months
  The bone around the implant will be radiographically evaluated in terms of possible resorption measured, using ImageJ software (NIH freeware), on the distal and mesial aspect of each implant at each time point where it is foreseen.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Alberto Valente, DDS, MS, PhD, Principal Investigator — University of Cagliari
Locations (1):
- Policlinico Duilio Casula, AOU Cagliari, Monserrato, CA, Italy